CLINICAL TRIAL: NCT05029661
Title: Ultrafast Ultrasonic COMpound Push Wave imAging and Strain eStimation (Ultra-COMPASS) for Individual Plaque Stratification in the Carotid Arteries
Brief Title: Ultrasound Elastography for Individual Carotid Plaque Stratification
Acronym: Ultra-COMPASS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL77726.091.21
Record Dates: First submitted 2021-08-19; First posted 2021-08-31 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2021-08

CONDITIONS: Carotid Artery Plaque
Keywords: Ultrasound; Shear wave elastrography; Lipid-lowering medication; Atherosclerotic plaques
MeSH Terms: conditions — Carotid Stenosis; Plaque, Atherosclerotic | interventions — Ultrasonography, Carotid Arteries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No intervention: No intervention
  Interventions: Diagnostic Test: Carotid ultrasound

INTERVENTIONS:
Diagnostic Test: Carotid ultrasound — * Ultra-COMPASS measurements (longitudinal + cross-sectional) Shear wave elastography: plaque stiffness Strain elastrogaphy: plaque deformation B-mode visualization: geometry
  * Intima-media thickness
  * Pulse wave velocity

SUMMARY:
Ischemic strokes are a leading cause of death and disability worldwide. In 20% of cases they are caused by the rupture of atherosclerotic plaques in carotid arteries. Risk estimation of plaque rupture is currently suboptimal. Although pathology studies have shown that plaque composition provides a better risk assessment (lipid-rich core with thin fibrous cap = high risk (unstable plaque); fibrous core and a thick fibrous cap = low risk (stable plaque)), plaque composition cannot be determined using imaging techniques, and can therefore not be assessed non-invasively. Ultrasound, which is already widely used in clinical practice to determine plaque geometry could be an optimal technique to determine plaque composition and monitor plaques in a large population, due to its low patient burden, relatively low cost and speed of measurement. However, using conventional ultrasound it is not possible to reliably determine plaque composition. However, this might be possible using newly developed ultrasound functionalities(shear wave and strain elastography) enabling tissue stiffness estimation. It is known that recurrence risk is greatest in the first week after a stroke or transient ischemic attack (TIA) and decreases afterwards, probably due to a stabilization of the plaque due to a change in composition. Additionally, lipid-lowering medication is known to further reduce the recurrence risk after such an event, probably due to an acceleration of the stabilization process of the plaque. In this study, the investigators want to investigate whether Ultra-COMPASS ultrasound measurements (a combination of shear wave and strain elastography and ultrafast compounding (a fast variant of standard anatomical ultrasound to determine plaque geometry)) could be used to determine changes in plaque composition after a stroke / TIA.

Primary objective:

Investigate whether it is possible to detect plaque stabilization, determined by plaque stiffness, after a brain infarction or transient ischemic attack with Ultra-COMPASS ultrasound measurements.

Secundary objectives:

* Determine the association between (changes in) Ultra-COMPASS measurements and the lipid-lowering drugs used 6 and 12 weeks after ischemic stroke.
* Determine the association between Ultra-COMPASS measurements and recurrent cardiovascular events (TIA / cerebral infarction / myocardial infarction/death) 6 and 12 weeks after ischemic stroke.
* Determine the association between Ultra-COMPASS measurements and (changes in) low-density lipoprotein levels 6 and 12 weeks after ischemic stroke (if known).

Study design:

This is a prospective, longitudinal, observational, single-center cohort study in patients after a cerebral infarction or TIA with stenosis of one / both carotid arteries of 30-70% that receive or start withcholesterol-lowering medication. Ultra-COMPASS measurements will be taken within 7 days after brain infarction/TIA and at 6 ± 1 and after 12 ± 1 weeks in both carotid arteries to see if plaques stabilize overtime and to what extent medication stimulates a beneficial change in plaque composition.

ELIGIBILITY:
Inclusion Criteria:

* Transient ischemic attack in anterior flow area (with diffusion restriction on DWI/ADC sequences of the cerebral MRI, corresponding to recent ischemia) or clinical diagnosis of brain infarction (cerebral CT for exclusion of brain haemorrhage)
* Opportunity to undergo Ultra-COMPASS ultrasound measurements ≤7 days after initiation of first clinical symptoms
* Stenosis 30-70% of carotid arteries based on clinically performed carotid ultrasound or thickening of at least 2mm on CT/MR scan
* ≥18 jaar
* Signed informed consent

Exclusion Criteria:

* Total occlusion common carotid artery or internal carotid artery
* Cardio-embolic nature of ischemic stroke (a.o. atrial fibrilation, valvular prothesis, endocarditis, recent myocardialinfarction)
* Restenosis after carotid endarterectomy
* Acute myocardial infarction
* Radiotherapy-induced carotid stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a transient ischemic attack (diffusion restriction on DWI/ADC sequences of the cerebral MRI, corresponding to recent ischemia) or brain infarction and a carotid atherosclerotic plaque with a stenosis of 30-70% of (one of both) carotid arteries that receive or start with lipid-lowering drugs
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Alterations in plaque composition | 6 and 12 weeks
  Change in plaque composition (= change in plaque stiffness) measured with Ultra-COMPASS measurements (i.e. shear wave and strain elastography and plaque geometry) in patients with and without a change in lipid-lowering medication regimen

SECONDARY OUTCOMES:
Recurrent cardiovascular events | up to 12 weeks after brain infarction/TIA
  Determine the association between Ultra-COMPASS measurements (i.e. shear wave and strain elastography and plaque geometry) and recurrent cardiovascular events (TIA / cerebral infarction / myocardial infarction / death due to cardiovascular disease)
Lipoprotein level effect | 6 and 12 weeks after ischemic stroke (if known).
  Determine the association between Ultra-COMPASS measurements (i.e. shear wave and strain elastography and plaque geometry) and (changes in) low-density lipoprotein levels (if known).

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided